CLINICAL TRIAL: NCT00747422
Title: Evaluation of the Effectiveness and Safety of the Ulthera™ System for the Treatment of Periorbital Wrinkles
Brief Title: Evaluation of the Effectiveness and Safety of the Ulthera™ System for the Treatment of Wrinkles Around the Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ULT-102
Record Dates: First submitted 2008-09-03; First posted 2008-09-05 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2012-10

CONDITIONS: Periorbital Wrinkles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental)
  Interventions: Device: Ulthera™ System

INTERVENTIONS:
Device: Ulthera™ System — ultrasound treatment

SUMMARY:
The purpose of this study is to look at how safe and effective the Ulthera ultrasound system is at reducing the appearance of wrinkles when used with subjects who have wrinkles around the eyes.

DETAILED DESCRIPTION:
The purpose of this prospective, multi-center, single treatment, clinical trial is to evaluate the effectiveness and safety of the Ulthera™ System for the non-invasive treatment of periorbital wrinkles and rhytids.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 40 to 70 years
* Subject in good health
* Desire improvement in periorbital wrinkles
* Subject provides informed consent and agrees to attend follow-up visits
* Subject signs a HIPPA authorization

Exclusion Criteria:

* Pregnant or lactating
* Has an active systemic or local skin disease that may alter wound healing
* Has significant scarring in test areas
* Has significant open facial wounds or lesions
* Has severe or cystic acne on the face
* Has a metal stent or implant in the face area
* Is a current smoker or has a history of smoking in last 10 years

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
reduction of periorbital wrinkles | 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Scripps Clinic Carmel Valley, Division of Laser and Cosmetic Dermatology, San Diego, California
  - Northwestern University Department of Dermatology, Chicago, Illinois
  - SkinCare Physicians, Chestnut Hill, Massachusetts
  - Zel Skin and Laser Specialists, Edina, Minnesota